CLINICAL TRIAL: NCT03331367
Title: Investigating and Characterizing the Immune Response to Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 18-01696; 18-01696 (Other: NYU Langone Institutional Review Board)
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Prostate Cancer
Keywords: Cryotherapy; Radiation; Prostatectomy; Immune Response
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This study involves four arms consisting of patients who have undergone either total cryotherapy, focal cryotherapy, Cyberknife SBRT or radical prostatectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Total Cyrotherapy of the Prostate (Active Comparator): Patients who will undergo total cryotherapy of the prostate will be evaluated for immune markers using a blood draw and urine sample collected at three timepoints (baseline, 2-3 weeks post cryotherapy, 3 months post cryotherapy)
  Interventions: Procedure: Blood draw; Procedure: Urine sample
- Focal Cryotherapy of the Prostate (Active Comparator): Patients who will undergo focal cryotherapy of the prostate will be evaluated for immune markers using a blood draw and urine sample collected at three timepoints (baseline, 2-3 weeks post cryotherapy, 3 months post cryotherapy)
  Interventions: Procedure: Blood draw; Procedure: Urine sample
- Cyberknife SBRT of the Prostate (Active Comparator): Patients who will undergo Cyberknife SBRT of the prostate will be evaluated for immune markers using a blood draw and urine sample collected at three timepoints (baseline, 2-3 weeks post Cyberknife, 3 months post Cyberknife)
  Interventions: Procedure: Blood draw; Procedure: Urine sample
- Radical Prostatectomy (Active Comparator): Patients who will undergo a radical prostatectomy will be evaluated for immune markers using a blood draw and urine sample collected at three timepoints (baseline, 2-3 weeks post surgery, 3 months post surgery)
  Interventions: Procedure: Blood draw; Procedure: Urine sample

INTERVENTIONS:
Procedure: Blood draw — Patients in all four study arms will provide a blood sample to evaluate the immune response to prostate cancer treatment.
Procedure: Urine sample — Patients in all four study arms will provide a urine sample to evaluate the immune response to prostate cancer treatment.

SUMMARY:
This study is a clinical study to investigate and characterize the immune response profile to four different prostate cancer treatments (total cryotherapy, focal cryotherapy, Cyberknife SBRT, and radical prostatectomy) in patients with localized prostate cancer.

DETAILED DESCRIPTION:
The immune system plays an important role in cancer, and there is evidence that different types of cancer treatment can elicit different responses from the body's immune system. This study is designed to look at immune markers in the blood and urine of patients undergoing four different types of prostate cancer treatment and compare the differences.

Patients who have elected Total Cryotherapy (freezing of the entire prostate), focal cryotherapy (freezing only the side of the prostate affected by cancer), Cyberknife stereotactic body radiation therapy (SBRT) and Radical Prostatectomy (removal of the entire prostate) for the treatment of their prostate cancer will be eligible to participate in this study. The study is expected to enroll 40 patients, 10 patients per treatment group. The study includes a screening visit during which the subject will provide informed consent, and provide a blood sample and a urine sample. At 2-3 weeks following their scheduled treatment, they will again provide another blood and urine sample. At their regularly scheduled follow up at 3 months, they will again provide another blood and urine sample. These samples are collected for research purposes only, and the costs will be covered by the study grant account, without any additional cost to the patient.

The investigators have determined that this study presents no more than minimal risk to patients due to the minimal risks involved with a blood draw and urine specimen collection.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to freely sign informed consent to enroll in the study.
* Histologically proven Prostate Carcinoma.
* Undergoing total cryotherapy, focal cryotherapy, Cyberknife SBRT or radical prostatectomy for prostate cancer treatment.

Exclusion Criteria:

* Has previously had a radical prostatectomy for prostate cancer.
* Has previously received cryotherapy for prostate cancer.
* Previous treatment with chemotherapy within the past 6 months.
* Previous treatment with radiation within the past 18 months.
* Has evidence of metastatic disease.
* Has a current or history within the past 6 months of alcohol and/or substance abuse which would impair participation in the study.
* Has a major medical disorder (i.e. uncontrolled diabetes, significant hepatic, renal or hematological disorders, recent stroke or myocardial infarction), in the opinion of the urologist, is an illness or complication which is not consistent with the protocol requirements.
* Is not willing to undergo the necessary follow-up for the trial period.
* Has known immunologic disease, human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Evaluate the change in blood cytokine profile | Before treatment, 2-3 weeks post treatment, 3 months post treatment
  Cytokines to be evaluated include but are not limited to: TNF-alpha, IL-1b, IL2, IL-2 CD25 Receptor Soluble, IFN-gamma, IL-4, IL-5, IL-6, IL-8, IL-10, IL-12 and IL-13.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron E Katz, MD, Principal Investigator — NYU
Locations (1):
- NYU Winthrop Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: No